CLINICAL TRIAL: NCT05304247
Title: Prevalence and Risk Factors of Black Tooth Stains and Their Relation With Caries Experience in Primary Teeth of A Group of Preschool Children: A Cross-Sectional Study.
Brief Title: Prevalence and Risk Factors of Black Tooth Stains
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mennatallah Hesham Elsayed Mohamed Ali (Other)
Responsible Party: Sponsor-Investigator, Mennatallah Hesham Elsayed Mohamed Ali, Principal investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: prevalence of BS
Record Dates: First submitted 2022-02-12; First posted 2022-03-31 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Dental Plaque
Keywords: black stains
MeSH Terms: conditions — Dental Plaque | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire and clinical examination — Prevalence and Risk Factors of Black Tooth Stains and Their Relation With Caries Experience in Primary Teeth of A Group of Preschool Children

SUMMARY:
To assess the prevalence of black tooth stains and their relation with caries experience in the primary dentition of 3-5-year-old children.

DETAILED DESCRIPTION:
Tooth discoloration is frequently seen by dental practitioners and is considered an aesthetic problem. There are two types of teeth discoloration; intrinsic discoloration which is related to intrinsic factors such as congenital and inherited conditions and extrinsic discoloration which occurs due to the formation of pigments on the enamel surface (Prskalo et al., 2017).

Black stain is a specific type of external tooth discoloration. It is clinically diagnosed as dark dots on the gingival third of the tooth that may coalesce and form a complete dark line following gingival contour or can also impregnate pits, fissures, and grooves (França-Pinto et al., 2012).

Black stains are a common finding in children and are seen equally in both genders (Zyła et al., 2015). When children's smiles do not fit the esthetic criteria, it can have negative social and psychological consequences causing embarrassing situations for the child, including school bullying. Their guardians may also be affected as people could judge it as bad oral health and question the care given to these children .(Fernando Pessoa, n.d.)

The etiology of black stains is multifactorial . Chromogenic anaerobic bacteria have been considered one of the etiological factors by their production of hydrogen sulfide that interacts with iron present in saliva and forms insoluble ferric sulfate which is the main component of these pigments (Elelmi et al., 2021).

Rational:

Although black stains have been considered a protective factor against caries, they are considered a common aesthetic problem. According to the systematic review of Asokan et al., 2020, there is conflicting data on the relation between tooth stains and dental caries as some studies showed a positive association between black stains and caries and other studies showed a negative association between them, and therefore, further studies are needed to completely understand the nature, risk factors of black stains and their relation with caries experience.

ELIGIBILITY:
Inclusion Criteria:

* • 3-5 years old preschool children

  * Children with primary dentition

Exclusion Criteria:

• Children whose parents refuse signing informed consent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A Group of Egyptian Preschool Children
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of black tooth stains | base line
  measurement method : clinical examination used to asses the prevalence of black stains . unit of measurement : binary ( yes , no ) .

SECONDARY OUTCOMES:
Risk factors of black tooth stains | base line
  measurement method : questionnaire used to asses the risk factors of black stains . unit of measurement : binary questions ( yes , no ) .
caries experience | base line
  measurement method : dmf caries index used to asses the caries experience ,unit of measurement : scores .

REFERENCES:
- [Background] Elelmi Y, Mabrouk R, Masmoudi F, Baaziz A, Maatouk F, Ghedira H. Black stain and dental caries in primary teeth of Tunisian preschool children. Eur Arch Paediatr Dent. 2021 Apr;22(2):235-240. doi: 10.1007/s40368-020-00549-3. Epub 2020 Jul 8. PMID 32643037
- [Background] Franca-Pinto CC, Cenci MS, Correa MB, Romano AR, Peres MA, Peres KG, Matijasevich A, Santos IS, Barros AJ, Demarco FF. Association between black stains and dental caries in primary teeth: findings from a Brazilian population-based birth cohort. Caries Res. 2012;46(2):170-6. doi: 10.1159/000337280. Epub 2012 Apr 6. PMID 22488298
- [Background] Asokan S, Varshini KR, Geetha Priya PR, Vijayasankari V. Association between black stains and early childhood caries - A systematic review. Indian J Dent Res. 2020 Nov-Dec;31(6):957-962. doi: 10.4103/ijdr.IJDR_327_20. PMID 33753668
- [Background] Fernando Pessoa, U. (n.d.). Blanche Delcourt Chromogenic bacteria in the oral cavity and social impact in pediatric dentistry-A Literature Review
- [Background] Prskalo K, Klaric Sever E, Aleric I, Antonic Jelic T, Zaja I. Risk Factors Associated with Black Tooth Stain. Acta Clin Croat. 2017 Mar;56(1):28-35. doi: 10.20471/acc.2017.56.01.05. PMID 29120125